CLINICAL TRIAL: NCT01273753
Title: Using Bioimpedance Analysis and Blood Volume Monitoring to Assess the Impact of Intradialytic Exercise
Brief Title: Effects of Intradialytic Exercise as Assessed by Bioimpedance Analysis and Blood Volume Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Principal Investigator, Michael Heung, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Heung-BIA1
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Kidney Failure, Chronic
Keywords: End-stage renal disease; Hemodialysis; Bioimpedance analysis; Blood volume monitoring
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Active Comparator): After baseline measurements, all subjects will undergo a phase involving intradialytic exercise. Subjects will serve as their own controls.
  Interventions: Other: Intradialytic exercise

INTERVENTIONS:
Other: Intradialytic exercise — Patients will exercise using a stationary foot pedal cycle for 20 minutes at the beginning of hemodialysis.

SUMMARY:
The purpose of this study is to examine the impact of exercise during dialysis using objective measures of fluid status determination, specifically bioimpedance analysis (BIA) and blood volume monitoring (BVM). We hypothesize that exercise during dialysis will be associated with more stable blood pressures and that this will be reflected in different output from BIA and BVM monitoring.

DETAILED DESCRIPTION:
Achieving dry weight (DW) is essential for the optimal health of dialysis patients. Despite being one of the most basic and important factors in the management of hemodialysis patients, there are many obstacles to achieving DW. One problem underlying optimal fluid status management lies in the clinical assessment used to determine DW. The current standard is clinical judgment which is often reactive (ie. setting a weight below which the patient develops hypotension or cramping) instead of goal directed (ie. trying to achieve defined target measures). Moreover, DW is a dynamic parameter that changes in patients over time, and ongoing assessment remains reactive to changes in clinical status instead of proactively based on monitoring of validated measures. A primary impediment to achieving DW is the relatively short time during dialysis limiting vascular refilling and leading to complications of hypotension and other adverse sequelae of relatively rapid volume removal. The evaluation of interventions aimed at improving symptoms and preventing complications will be scientifically strengthened by objective assessment of the patient's volume. Fortunately two objective clinically validated tools to assess volume status have emerged: bioimpedance (BIA) which allows assessment of the patient's hydration status and blood volume monitoring (BVM) which allows direct measure of the rate of vascular refilling during dialysis. These will be essential in understanding the impact of therapeutic interventions directed at improving achievement of DW.

The next important consideration is selecting an intervention that shows promise in assisting patients in achieving DW. While many interventions deserve careful analysis we select exercise because of the additional cardiovascular benefits of exercise, and it fits into our outpatient program as part of achieving our overall outpatient wellness objectives. To this end we propose the following specific aim:

Specific Aim: Systematically evaluate the effects of exercise on hemodynamic stability and achievement of dry weight by testing the following hypotheses.

Hypothesis 1: Exercise bike riding during dialysis improves vascular refilling as determined by BVM.

Hypothesis 2: Exercise bike riding during dialysis improves (leads to a reduction in) tissue hydration status as determined by BIA.

Hypothesis 3: Improved intra-dialytic blood pressure stability is directly related to improved vascular refilling as assessed by BVM, which is in turn related to improved (reduced) tissue hydration as assessed by BIA.

Hypothesis 4: Intravascular refilling (assessed by BVM) is directly related to reduction in tissue hydration (assess by BIA).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18yrs and older
2. End-stage renal disease on thrice weekly maintenance hemodialysis for at least 3 months
3. Stable dry weight for the preceding month
4. Stable dialysis prescription for the preceding month
5. Average interdialytic weight gain at least 1kg but less than 4% of total body weight.

Exclusion Criteria:

1. Patients receiving dialysis for acute renal failure
2. Hospitalization >1 day in the preceding month
3. Inability to complete exercise regimen or medical contraindication to exercise regimen
4. Patients in whom a dry weight is yet to be established
5. History of non-compliance with dialysis therapy (defined as > 3 missed treatments in a month)
6. Inability to remain in horizontal position for duration of a dialysis session.
7. Amputation of a limb other than fingers or toes.
8. Pace maker, defibrillator, implantable pump, artificial joint, pins, plates or other types of metal objects in the body (other than dental fillings).
9. Coronary stents or metal suture material in the heart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in bioimpedance analysis trend during dialysis | Baseline (no exercise) and 4 weeks (with exercise)
  The investigators will assess the impact of intradialytic exercise on body composition and fluid removal by comparing BIA measurements and trends between dialysis treatments. The baseline measurement will occur during standard usual dialysis, while the 4 week meaurement will occur during dialysis with exercise.

SECONDARY OUTCOMES:
Blood volume monitoring | Baseline (no exercise) and 4 weeks (with exercise)
  Blood volume monitoring will be done during dialysis to assess the impact of exercise on the slope of blood volume changes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Heung, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States